CLINICAL TRIAL: NCT00610077
Title: An Open, Randomized, Parallel-Group, Multicentric, Comparative Study of Letrozole With Clomiphene Citrate for Induction of Ovulation in Anovulatory Infertility.
Brief Title: Letrozole vs. Clomiphene Citrate in Patients With Anovulatory Infertility
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Medical Advisor, Sun Pharmaceutical Industries Limited
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LET/SPIL/03/06
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Last update posted 2008-02-07 (Estimated); Status verified 2008-01

CONDITIONS: Infertility
Keywords: Letrozole; Clomiphene citrate; Anovulatory infertility; Ovulation induction
MeSH Terms: conditions — Infertility | interventions — Letrozole; Clomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Letrozole
  Interventions: Drug: Letrozole
- 2 (Active Comparator): Clomiphene citrate
  Interventions: Drug: Clomiphene citrate

INTERVENTIONS:
Drug: Letrozole — Tablet Letrozole 2.5 mg once a day for 5 days for 3 cycles
  Other Names: Letroz
  Arms: 1
Drug: Clomiphene citrate — Clomiphene citrate 100 mg or 150 mg once a day for 5 days in 3 cycles
  Other Names: Ferotab
  Arms: 2

SUMMARY:
OBJECTIVE: To compare the effectiveness of letrozole and clomiphene citrate (CC) in patients with anovulatory infertility. DESIGN: Open, prospective, randomized, parallel group, multicentric, comparative trial. SETTING: Out patient clinics of infertility centers in India. PATIENT(S): Fifty-five patients with anovulatory infertility were recruited. Twenty-seven patients (59 cycles) were given letrozole and twenty-eight patients (68 cycles) were given CC. Both drugs were given orally on days 3-7 of menstrual cycle. INTERVENTION(S): Letrozole, CC, ovulation induction, vaginal micronized progesterone, IUI.

DETAILED DESCRIPTION:
MAIN OUTCOME MEASURE(S): Occurrence of ovulation, endometrial thickness and pregnancy rates.

ELIGIBILITY:
Inclusion Criteria:

* Females with anovulatory infertility 20-38 years of age.
* Diagnosis of anovulatory infertility as established by standard criteria.
* Normal Pelvic USG and bilateral tubal patency
* Willingness and giving written Informed Consent.

Exclusion Criteria:

* Uterine and adnexal pathology e.g. leiomyomata
* Ovarian cyst
* Hyperprolactinaemia
* Hyperthyroidism or Hypothyroidism*
* FSH >9mIU/ml (during early follicular phase).* (As per Chemoluminescence method)
* Previous surgery related to genital tract as per history
* Appendicitis, peritonitis, genital tuberculosis as per history and/or having an abnormal pelvic anatomy
* Impaired hepatic /renal function
* Diabetes mellitus/Random blood sugar- > 140mg/dl
* Drugs likely to interfere with ovulation
* Alcohol intake as per history
* History of hypersensitivity to the study drug or to its excipients
* Planned travel outside the study area for a substantial portion (>5 days) of the study period by potential participants
* Lack of willingness to give informed written consent
* Participation in any clinical study within the preceding 1 month

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2004-12; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Ovulation rate (ovulatory cycles/ all treatment cycles) by Ultrasonography (USG). | 3 cycles

SECONDARY OUTCOMES:
Pregnancy Rate (Detection of pregnancy by beta-hCG and Ultrasonography) b. Endometrial thickness by Ultrasonography. | 3 cycles
Safety | 3 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Mandakini Parihar, M.D., D.G.O., Principal Investigator — Director, IVF Centre, Chembur
Locations (1):
- IVF Centre, Chembur,, Mumbai, Maharashtra, India